CLINICAL TRIAL: NCT06327984
Title: Barts Sex-CAD Database: Do Female Sex Hormone Levels Inform Inflammatory Status and Susceptibility in Women Suffering Coronary Artery Disease?
Brief Title: Barts Sex-CAD Database - Sex Hormones and Inflammatory Status in Coronary Artery Disease
Status: Recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 157354
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Acute Coronary Syndrome; Atherosclerosis; Inflammation
Keywords: Coronary artery disease; Acute coronary syndrome; Myocardial infarction; Sex characteristics; Hormones; Inflammation
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Acute Coronary Syndrome; Atherosclerosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Plasma samples from human blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a lack of understanding of how Coronary Artery Disease (CAD) - meaning the blocking or furring up of the arteries of the heart - starts and progresses in women. In both men and women, CAD is the most common cause of heart attacks, which occur when the blood supply in the heart is interrupted (these are also known medically as 'acute coronary syndromes').

Before the menopause women appear to be protected from CAD; however, after the menopause that protection is lost. Also, those women who do suffer a heart attack have twice the risk of further heart attacks compared to men despite having the same treatment that works well in men. Biological differences between men and women are probably playing an important role in the way CAD develops. However, due to a lack of research there is currently little understanding of how the female body works in this area.

Inflammation is the body's natural response to injury or infection. Importantly it is also involved in the development of CAD. Hormones such as oestrogen and testosterone are also likely to be contributory factors. The investigators think the differences between the way these hormones and inflammation play a part in CAD in both men and women are important, but the role they play is not yet fully understood.

In this study the investigators wish to measure the 'markers' of inflammation in the blood of patients attending Barts Heart Centre with chest pain. The investigators will also conduct questionnaires with these patients, to understand their hormone status and how parts of their medical history may be a contributory factor. For patients who have previously attended Barts Heart Centre will will contact them to conduct the questionnaire over the telephone only. The investigators will combine this data with the data that is routinely collected during hospital admission. In this way the investigators hope to understand whether inflammation together with hormone status plays an important role in CAD. Our hope is that through this research the investigators will address an under researched area and find new ways of treating women and men with coronary artery disease.

DETAILED DESCRIPTION:
1. The investigators will collect data on sex hormone status (FSH, LH, oestradiol, progesterone and testosterone) of patients admitted to BHC. Data will subsequently be entered into a dedicated secure database by a member of the clinical team. A member of the clinical team will review hormone profiles and, if relevant abnormalities in hormone profiles are detected, appropriate follow up will be arranged for the patient. In addition, the following blood markers will also be extracted from the patients routine admission blood tests: Haemoglobin, white blood cell count, platelet count, haematocrit, neutrophil count, lymphocyte count, monocyte count, eosinophil count, coagulation results, d-dimer (if done), sodium, potassium, chloride, urea, creatinine, eGFR, bilirubin, ALT, ALP, protein, albumin, calcium, corrected calcium, phosphate, magnesium, troponin, hs-CRP. These data points will be logged in the secure database.
2. We have composed a short questionnaire to examine aspects of patients' history relevant to their sex hormone status. For female patients this includes menstrual history, as well as relevant medications and medical conditions that may influence sex hormone status. For males an abbreviated form of the questionnaire includes relevant medications and medical conditions that my influence sex hormone status. This questionnaire will be delivered retrospectively to patients following their discharge from hospital. Clinical data has been gathered into the BartsREVASC database since 2016 therefore we aim to retrospectively include these patients and contact them via telephone to conduct the questionnaire only. Patients will be identified via the BartsREVASC database, and the electronic patient record and NHS Spine record will be checked to ensure the patient is still living and has appropriate capacity to consent. An text message will be sent to retrospective patients with provides a link to the study information and invitation letter which will advise that they will receive a phone call from a clinical member of the research team to conduct the questionnaire over the telephone. A telephone number for the research team will be provided if they wish to call us sooner at their own convenience to conduct the questionnaire rather than receive a call. We will obtain their verbal consent (which will be documented in a database) prior to proceeding with the questionnaire; data will be directly entered into the secure database. Questionnaires will be administered by a member of the clinical team who will also be responsible for entering the data into the database. In addition, we will consent patients to be contacted regarding future research studies examining sex differences in CAD and inflammation.
3. Will seek also written consent from female and male patients prospectively included in this study during their hospital admission to obtain an additional blood test for specialised inflammatory profiling including but not limited to inflammatory cell count, white blood cell activation markers, markers of apoptosis, markers of cell death, inflammatory cytokine levels. These blood samples will be analysed at the William Harvey Research Institute, Queen Mary University of London using standard laboratory techniques. The investigators will also seek written consent from these patients to take part in the questionnaires outlined above for females and males. The questionnaires will be delivered in person at the time of blood sampling or over the telephone after discharge. In addition, the investigators will consent patients to be contacted regarding future research studies examining sex differences in CAD and inflammation. All data will be added to the secure database.
4. In the circumstance where additional blood tests reveal significant results that require action. The investigators will inform the patient and the patients direct care team if applicable (e.g for current inpatients). If necessary, a referral to an appropriate specialist will be done with the patients consent. The investigators will also write to the patients' general practitioner in this circumstance to inform them of the results and action performed or required.
5. Novel data held in the secure database will be cross analysed with routine clinical data from the BartsREVASC database, electronic patient record and other relevant databases if required such as the MINOCA database in order to establish relationships,for follow up and MACE outcome data (see below),. Protecting patient's data is important and therefore data will be pseudonymised before being used for research purposes.
6. Patients will be followed up at 30 days/1 year/5years using electronic patient records at to determine outcomes including but not limited to medication data, all-cause mortality, readmission rates and further cardiovascular events.

ELIGIBILITY:
Inclusion criteria Any patient presenting with chest pain ≥16 years old presenting to Barts Heart Centre will be included.

Exclusion criteria Patients <16 years old and Adults lacking capacity will be excluded. Patients where the cause of their chest pain presentation is not related to coronary artery disease e.g musculoskeletal chest pain, aortic dissection, gastrointestinal, pulmonary embolism

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients attending Barts Heart Centre with chest pain
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2033-01-31 (Estimated); Study Completion 2033-01-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days/1 year/5 years
  Mortality at 30 days,1 year and 5 years, and relation to sex hormone/menstrual status/inflammatory profile
Re-admission | 30 days/1 year/5 years
  Re-admission rates post revascularization and relation to sex hormone/menstrual status/inflammatory profile
MACE | 30 days/1 year/5 years
  MACE post revascularisation and relation to sex hormone/menstrual status/inflammatory profile

SECONDARY OUTCOMES:
Relationship with specific MI types | 30 days/1 year/5 years
  Relationship of sex hormone/menstrual status/inflammatory profile with specific types of ACS such as MINOCA
Relationship with inflammation | 30 days/1 year/5 years
  Relationship of sex hormone/menstrual status with markers of inflammation (e.g white cell count, CRP, D-dimer) and severity of disease (e.g troponin, extent of coronary disease)

CONTACTS AND LOCATIONS:
Overall Officials: Krishnaraj Rathod, MBBS PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee MT, Mahtta D, Ramsey DJ, Liu J, Misra A, Nasir K, Samad Z, Itchhaporia D, Khan SU, Schofield RS, Ballantyne CM, Petersen LA, Virani SS. Sex-Related Disparities in Cardiovascular Health Care Among Patients With Premature Atherosclerotic Cardiovascular Disease. JAMA Cardiol. 2021 Jul 1;6(7):782-790. doi: 10.1001/jamacardio.2021.0683. PMID 33881448
- [Background] Shabbir A, Rathod KS, Khambata RS, Ahluwalia A. Sex Differences in the Inflammatory Response: Pharmacological Opportunities for Therapeutics for Coronary Artery Disease. Annu Rev Pharmacol Toxicol. 2021 Jan 6;61:333-359. doi: 10.1146/annurev-pharmtox-010919-023229. Epub 2020 Oct 9. PMID 33035428
- [Result] Rathod KS, Jones DA, Jain AK, Lim P, MacCarthy PA, Rakhit R, Lockie T, Kalra S, Dalby MC, Malik IS, Whitbread M, Firoozi S, Bogle R, Redwood S, Cooper J, Gupta A, Lansky A, Wragg A, Mathur A, Ahluwalia A. The influence of biological age and sex on long-term outcome after percutaneous coronary intervention for ST-elevation myocardial infarction. Am J Cardiovasc Dis. 2021 Oct 25;11(5):659-678. eCollection 2021. PMID 34849299